CLINICAL TRIAL: NCT01176916
Title: A PROSPECTIVE PRAGMATIC CLINICAL TRIAL OF CHINA EARLY INVASIVE BREAST CANCER PATIENTS RECEIVING ADJUVANT THERAPY WITH AROMASIN
Brief Title: Aromasin® Interventional Study Of Early Invasive Breast Cancer Patients In China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None
Other Study IDs: A5991093; NRA5990043 (Other: Alias Study Number)
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; Aromasin; adjuvant chemotherapy; endocrine therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Aromasin (exemestane)

INTERVENTIONS:
Drug: Aromasin (exemestane) — the dosage, frequency and duration base on the LPD approved by SFDA.

SUMMARY:
Aromasin® (Exemestane) was approved in China for adjuvant treatment of postmenopausal women with estrogen receptor (ER) positive early invasive breast cancer who have received 2-3 years of tamoxifen & are switched to Aromasin® for completion of a total of 5 consecutive years of adjuvant hormonal therapy by State Food and Drug Administration (SFDA) with clinical trial waive. While Aromasin® has been used in China for adjuvant therapy of breast cancer since then, there is currently lack of systematic collection and analysis for the efficacy and safety data of Aromasin® adjuvant setting in Chinese population. The Aromasin® Interventional Study is being proposed to collect data systematically and to assess the efficacy and safety of Aromasin® adjuvant setting in Chinese population.

DETAILED DESCRIPTION:
This is interventional study and single arm study. N/A

ELIGIBILITY:
Inclusion Criteria:

* Early invasive breast cancer (T1-4N1-3M0) confirmed by histology or cytology.
* ER positive.
* The patient must be postmenopausal woman.
* The patient has received adjuvant Tamoxifen therapy for up to 2-3 years and will switch to receive Aromasin® treatment (The decision to prescribe Aromasin® will necessarily precede and will be independent of the decision to enroll patients in the study).

Exclusion Criteria:

* Following the adjuvant Tamoxifen therapy for 2-3 years and prior to receiving Aromasin® treatment, there is evidence of a local relapse or distant metastasis of breast cancer, or a second primary cancer.
* Following the adjuvant Tamoxifen therapy for 2-3 years and received other aromatase inhibitors (not Aromasin®).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The patient must be postmenopausal woman.
Enrollment: 564 (Actual)
Dates: Start 2011-02-09 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- China (53):
  - The First Affiliated Hospital of Bengbu Medical College/Medical Oncology Department, Bengbu, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Second Affiliated hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First hospital of LanZhou university, Lanzhou, Gansu
  - Breast Surgery of The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - SUN YAT-SEN Memorial Hospital , SUN YAT-SEN University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Thyroid and breast surgery, Shenzhen, Guangdong
  - Affiliated hospital of Guangdong medical college, Zhanjiang, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Weihui, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan provincial people's hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Jingzhou Hospital Tongji Medical College Huazhong university of science and Technology, Jingzhou, Hubei
  - Breast and thyroid surgery of the Central Hospital of WuHan, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University /Department of Breast, Changsha, Hunan
  - The Affiliated Hospital of inner Mongolia medical university, Hohhot, Inner Mongolia
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Jiangsu Cancer Hospital/ Surgery Department, Nanjing, Jiangsu
  - Jinling Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital/ Surgery Department, Nanjing, Jiangsu
  - Nanjing Maternity and Child Health Care Hospital/Department of Breast Surgery, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - The first hospital of jilin university, Changchun, Jilin
  - The Fourth Affiliated Hospital Of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of The Fourth Military Medical University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Linyi People's Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Qingdao municipal Hospital, Qingdao, Shandong
  - Breast Surgery of The Weifang People's Hospital, Weifang, Shandong
  - Breast Surgery of YanTai Yu Huang Ding Hospital, Yantai, Shandong
  - Breast and thyroid surgery of Central Hospital of Zibo, Zibo, Shandong
  - West China Hospital, Sichuan University/ Oncology Department, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin Cancer Hospital/Breast cancer department, Tianjin, Tianjin Municipality
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Cancer Hospital Chinese Academy of medical sciences, Beijing
  - Fifth Medical Center of the PLA General Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital/Department of Oncology, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Fudan University Shanghai Cancer center/Department of Breast Surgery, Shanghai
  - Yangpu District Central Hospital, Shanghai
  - Xinhua Hospital Affiliated to Shanghai JiaoTong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 564 participants were assigned into the study and 558 participants received the study treatment. (6 participants were withdrawn from the study prior to the first dose of Aromasin.)
Groups:
- Exemestane: Participants received exemestane (Aromasin) tablet 25 mg once daily in this study. They had previously taken tamoxifen for 2 to 3 years and switched to Aromisin in this study for completion of 5 consecutive years of adjuvant hormonal therapy.
Period: Overall Study
Arm/Group | Exemestane
Started | 564
Treated | 558
Assigne But Not Treated | 6
Completed | 397
Not Completed | 167
Not completed — Adverse Event | 61
Not completed — Death | 1
Not completed — Lost to Follow-up | 15
Not completed — Objective progression or relapse | 17
Not completed — Protocol Violation | 24
Not completed — Withdrawal by Subject | 37
Not completed — Other | 6
Not completed — Withdrawal prior to Treatment | 6

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who were treated.
Arm/Group | Exemestane
Number analyzed (Participants) | 558
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 558
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 558
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Time-to-Event
Description: An event was defined as the earliest occurrence of any of the following: 1) Loco-regional/distant recurrence of the primary breast cancer (BC) (Loco-regional recurrence was defined as any recurrence in the ipsilateral breast, chest wall or axillary lymph nodes.); 2) Appearance of a second primary or contralateral breast cancer; 3) Death due to any cause.
Time Frame: 2-3 years (time for previously taking tamoxifen [prior to this study] and time for taking Aromasin [in this study] add up to 5 years)
Population: The full analysis set (FAS) was defined as all participants who received at least 1 dose of Aromasin during the observation period. All efficacy analyses were performed using the FAS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Exemestane
Number analyzed (Participants) | 558
months | NA [NA to NA] — The median (95% confidence interval [CI]) time to event was not estimable because only a small number of participants experienced the event by the end of study.

2. Secondary Outcome: Percentage of Participants Experiencing Each Event
Description: An event was defined as the following: 1) Loco-regional/distant recurrence of the primary breast cancer (Loco-regional recurrence was defined as any recurrence in the ipsilateral breast, chest wall or axillary lymph nodes.); 2) Appearance of a second primary or contralateral breast cancer; 3) Death due to any cause.
Time Frame: as for outcome 1
Population: The FAS was defined as all participants who received at least 1 dose of Aromasin during the observation period. All efficacy analyses were performed using the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Exemestane
Number analyzed (Participants) | 558
percentage of participants
  Loco/distant recurrence of the primary BC | 3.0 [1.91 to 4.82]
  Second primary/contralateral BC | 0.4 [0.10 to 1.30]
  Death due to any cause | 0.7 [0.28 to 1.83]

3. Secondary Outcome: Incidence Rate of Each Event
Description: Incidence rate (per annum) of the event was defined as a ratio of the number of events and the total exposure time (in years) to Aromasin therapy.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: events per person-year
Arm/Group | Exemestane
Number analyzed (Participants) | 558
events per person-year
  Loco/distant recurrence of the primary BC | 0.02995
  Second primary/contralateral BC | 0.00352
  Death due to any cause | 0.00321

4. Secondary Outcome: Hazard Ratio: the Relationship Between (Human Epidermal Growth Factor Receptor 2) HER2 Status and Time-to-Event
Description: A Cox proportional hazards regression model was used to evaluate the relationship between HER2 status level (binary) and time-to-event (Positive vs Negative). The method for selecting factors for the Cox regression model was based on significant results at univariate analysis and the clinical judgement for the multivariate model. Stepwise method was used for the selection of final independent variables. The criteria for stepwise selection were pentry = 0.25 and pstay = 0.15.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Exemestane
Number analyzed (Participants) | 558
ratio | 0.835 [0.274 to 2.542]

5. Secondary Outcome: Harzard Ratio: the Relationship Between Multiple Disease Variables and Time-to-Event
Description: A Cox proportional hazards regression model with stepwise selection was used to evaluate the influence of multiple disease variables on the time-to-event. The disease variables in the initial model included Eastern Cooperative Oncology Group [ECOG] performance status at diagnosis; and Tumor, Lymph Node and Metastasis [TNM] stage at initial diagnosis. The ECOG Performance Status describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability. ECOG performance status at diagnosis level included 0, 1, 2, 3 and 4, with Level 0 as the best status and Level 4 as the worst. The TNM system helps describe the size of cancer tumor and the extent to which it spreads to nearby tissues/distant parts of the body. TNM stage at initial diagnosis level included 1 (Stage I), 2 (Stage IIA), 3 (Stage IIB), 4 (Stage IIIA), 5 (Stage IIIB) and 6 (Stage IIIC), with Level 1 as the best status and Level 6 as the worst.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Exemestane
Number analyzed (Participants) | 558
ratio
  ECOG performance status at diagnosis | 2.079 [0.773 to 5.591]
  TNM stage at initial diagnosis: number analyzed (Participants) | 532
  TNM stage at initial diagnosis | 1.532 [1.129 to 2.080]

6. Secondary Outcome: Number of Participants With Discontinuation Due to Adverse Events (AEs)
Description: Participants permanently discontinued from the study due to AEs were counted for this outcome measure. An AE is any untoward medical occurrence in a clinical investigation subject administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. The number of participants with discontinuation due to all-causality and treatment-related AEs are reported below. Treatment-related AEs were determined by the investigator.
Time Frame: as for outcome 1
Population: The safety analysis set (SAS) was defined as all enrolled participants who took at least 1 dose of the study drug. All safety analyses were reported within the SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Exemestane
Number analyzed (Participants) | 558
Participants
  all-causality | 62
  treatment-related | 47

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: All-causality TEAEs were counted for this outcome measure. TEAE is defined as an event that emerges during treatment, having been absent pretreatment, or worsens relative to the pretreatment state. The number of participants with all-causality and treatment-related TEAEs are reported below. Treatment-related TEAEs were determined by the investigator.
Time Frame: as for outcome 1
Population: The SAS was defined as all enrolled participants who took at least 1 dose of the study drug. All safety analyses were reported within the SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Exemestane
Number analyzed (Participants) | 558
Participants
  all-causality | 345
  treatment-related | 222

ADVERSE EVENTS:
Time Frame: 2-3 years (time for previously taking tamoxifen [prior to this study] and time for taking Aromasin [in this study] add up to 5 years)
Description: The same event may appear as both an AE and a SAE. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Exemestane
All-Cause Mortality (participants affected / at risk) | 4/558
Serious Adverse Events (participants affected / at risk) | 38/558
Other Adverse Events (participants affected / at risk) | 82/558
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exemestane (N=558)
Angina unstable (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Tongue haemorrhage (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Localised infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Breast fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ewing's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral infarction (Nervous system disorders) | 4 (4)
Post herpetic neuralgia (Nervous system disorders) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Breast calcifications (Reproductive system and breast disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exemestane (N=558)
Arthralgia (Musculoskeletal and connective tissue disorders) | 50 (51)
Vaginal haemorrhage (Reproductive system and breast disorders) | 33 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT01176916/Prot_001.pdf
  • Statistical Analysis Plan (2015-06-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT01176916/SAP_000.pdf